CLINICAL TRIAL: NCT06516523
Title: Impact of Pulsed Electromagnetic Field (PEMF) on Human Peri-implant Tissues: Clinical, Proteomic Profile, and Histological Analysis of a Randomized Clinical Trial
Brief Title: Impact of Pulsed Electromagnetic Field (PEMF) on Human Peri-implant Tissues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guarulhos (Other)
Responsible Party: Principal Investigator, Jamil awad shibli, Professor, University of Guarulhos
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 52969221.0.0000.5193
Record Dates: First submitted 2024-07-17; First posted 2024-07-24 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Periodontitis; Dental Plaque
MeSH Terms: conditions — Periodontitis; Dental Plaque | interventions — Bone Regeneration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PEMF and Bone Formation (Experimental): Use of activated miniaturized device with PEMF
  Interventions: Procedure: PEMF and Control/Sham; Device: PEMF and without PEMF
- Control SHAM PEMF (Placebo Comparator): Use of SHAM miniaturized device with PEMF (without Pulse)
  Interventions: Procedure: PEMF and Control/Sham; Device: PEMF and without PEMF
- Non-surgical treament of peri-implantitis with PEMF (Active Comparator): USE of PEMF on the microbiome modulation and bone formation under inflammatory conditions
  Interventions: Procedure: PEMF and Control/Sham; Device: PEMF and without PEMF
- Non-surgical treatment of peri-implantitis without PEMF (Placebo Comparator): USE of SHAM (no PEMF) on the microbiome modulation and bone formation under inflammatory conditions
  Interventions: Procedure: PEMF and Control/Sham; Device: PEMF and without PEMF

INTERVENTIONS:
Procedure: PEMF and Control/Sham — Use o PEMF on test implants (treatment of peri-implantitis and bone formation) Use of PEMF on experimental implants (Bone-to-implant contact)
  Other Names: Bone regeneration; Treatment of peri-implantitis
Device: PEMF and without PEMF — Use o PEMF on test implants (treatment of peri-implantitis and bone formation)
  Other Names: Treatment of peri-implantitis

SUMMARY:
Pulsed Electromagnetic field (PEMF) has been shown to heighten bone regeneration and wound healing in various clinical areas, including dentistry. In Oral implantology, PEMF stimulation may enhance peri-implant bone formation and secondary stability and modulate the peri-implant microbiome. This randomized controlled study will evaluate:

1. the impact of PEMF around interim additive manufacturing (AM) implants immediately loaded and retrieved from human jaws after 60 days.
2. the effect of PEMF on diseased dental implants using non-surgical therapy.

DETAILED DESCRIPTION:
Non-surgical treatment of peri-implantitis:This is a prospective, double-blind, randomized, sham-controlled pilot study of a 3-month duration, as shown in the study flow chart (Figure 1). The data are reported according to the Consolidated Standards of Reporting Trials (CONSORT) guidelines. Treatment allocation was by block randomization, with a block size of four. Both patients and evaluators were blind to whether the MED device was active or not.

Patients who were diagnosed with peri-implantitis and fit the inclusion criteria were identified from the records. The inclusion criteria were: patients aged 20-85 years with evidence of peri-implant crestal bone loss greater than 3mm but not more than 5mm; presence of bleeding on probing or suppuration; an implant pocket depth of 6-8 mm; implants with an internal hex connection of 3.75-4.1mm diameter; implant-supported restoration that could be removed and later refitted; and patients who adhered to their scheduled periodontal maintenance visits. All patients in the study were under strict periodontal maintenance with no residual pockets at other sites at the time of diagnosis. Furthermore, all patients included in the study had signed an informed consent form.

Exclusion criteria were identified based on patient records and included: patients consuming medications that might affect soft and hard tissue healing/health (such as calcium channel blockers, immunosuppressive, and anticonvulsive medications); patients currently taking systemic antibiotics; chronic use of nonsteroidal anti-inflammatory drugs (NSAIDs) on a long-term basis (excluding low dose aspirin); presence of a pacemaker; patients with periodontal disease; cigarette smoking of more than 10 cigarettes a day; and missing data in patient's files.

Bone formation:The present study will be designed as a randomized controlled investigation, reporting on immediately loaded transitional transmucosal implants placed in the human posterior jaws and retrieved after 60 days. This study aims to compare the early peri-implant tissues response to implants with or without PEMF activation when placed in the human posterior jaws and subjected to immediate loading protocol. During a routine surgical procedure for the placement of conventional implants, each enrolled patient also will receive two transitional transmucosal implants (test-with and control-without PEMF), which were inserted in the posterior area of the jaws (mandible and maxilla), according to a randomization process. The transitional implants (3.0 mm x 10mm) will be placed to support an interim prosthesis until healing of the conventional implants. After 8 weeks, during the second-stage surgery to uncover the conventional implants, all transitional implants, and surrounding tissues will be retrieved for evaluation. This protocol was elaborated according to the Standard Protocol Items: Recommendations for Interventional Studies (SPIRIT) protocol. All eligible volunteers will be informed about the nature, potential risks, and benefits of participating in this study and will sign a free and informed consent term.

ELIGIBILITY:
Inclusion Criteria:

Bone formation

* good systemic and oral health
* sufficient native bone to place implants of 3.0 mm diameter and 10 mm length for the bone formation arm

treatment of peri-implantitis

* patients aged 18-85 years with evidence of peri-implant crestal bone loss greater than 3mm but not more than 5mm;
* the presence of bleeding on probing or suppuration;
* an implant pocket depth of 6-8 mm;
* implants with an internal hex connection of 3.75-4.1mm diameter;
* implant-supported restoration that could be removed and later refitted
* patients who adhered to their scheduled periodontal maintenance visits.

Exclusion Criteria:

* patients consuming medications that might affect soft and hard tissue healing/health (such as calcium channel blockers, immunosuppressive, and anticonvulsive medications)
* patients currently taking systemic antibiotics
* chronic use of nonsteroidal anti-inflammatory drugs (NSAIDs) on a long-term basis (excluding low dose aspirin);
* presence of a pacemaker; patients with periodontal disease;
* cigarette smoking of more than 10 cigarettes a day
* missing data in patient's files.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Non-surgical Treatment of peri-implantitis | 12 months
  reduction of probing depth
Bone formations under PEMF | 2 months
  BIC% increase

CONTACTS AND LOCATIONS:
Overall Officials: Jamil Shibli, Principal Investigator — Guaurlhos University
Locations (1):
- Guarulhos University, Guarulhos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faveri M, Miquelleto DEC, Bueno-Silva B, Pingueiro JMS, Figueiredo LC, Dolkart O, Yakobson E, Barak S, Feres M, Shibli JA. Antimicrobial effects of a pulsed electromagnetic field: an in vitro polymicrobial periodontal subgingival biofilm model. Biofouling. 2020 Aug;36(7):862-869. doi: 10.1080/08927014.2020.1825694. Epub 2020 Sep 29. PMID 32993357